CLINICAL TRIAL: NCT00002555
Title: A PHASE III RANDOMIZED STUDY ON POSTOPERATIVE RADIO- AND CHEMOTHERAPY IN PATIENTS WITH LOCALLY ADVANCED HEAD AND NECK CARCINOMAS
Brief Title: High-Dose Radiation Therapy With or Without Chemotherapy in Treating Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22931; EORTC-22931
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin

INTERVENTIONS:
Drug: cisplatin
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if radiation therapy plus chemotherapy is more effective than radiation therapy alone in treating patients with head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of high-dose radiation therapy alone with high-dose radiation therapy plus cisplatin in treating patients with head and neck cancer who have undergone surgery to remove the cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of cisplatin to high-dose postoperative radiotherapy increases the disease-free survival rate of patients with locally advanced head and neck carcinomas at high risk of recurrence following radical surgery.

OUTLINE: Randomized study. Patients are registered and randomized to treatment within 25 days of surgery. Arm I: Radiotherapy. Irradiation of the preoperative primary tumor site with a boost to areas at high risk for recurrence using Co60 equipment, 4-6 MV linear accelerators, or 6-12 MeV electrons. Arm II: Radiotherapy plus Single-Agent Chemotherapy. Irradiation as in Arm I; plus Cisplatin, CDDP, NSC-119875.

PROJECTED ACCRUAL: A total of 338 evaluable patients will be studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the head and neck of the following sites: Oral cavity Oropharynx Hypopharynx (only if ineligible for protocol EORTC-24891) Larynx T3-4, any N, M0 or any T, N2-3, M0 disease (UICC staging) resected with curative intent T3, N0 carcinoma of the larynx with suitable microscopically clear margins is ineligible At least one of the following high-risk characteristics required: Histopathologically positive surgical margins No gross residual disease Perineural involvement Extranodal spread of disease Oral cavity or oropharyngeal lesions with metastatic nodes at level 4 or 5 Vascular embolisms in the neck No metastases at diagnosis No known CNS disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-2 Hematopoietic: WBC at least 4,000 Platelets at least 100,000 Hemoglobin normal (at least 6.8 mmoles/liter) Hepatic: Bilirubin no greater than 2 times normal Other liver function tests no greater than 2 times normal Renal: Creatinine no greater than 1.3 mg/dL (120 micromoles/liter) Creatinine clearance greater than 60 mL/min Other: No active, uncontrolled infection No requirement for antibiotics that might interfere with platinum excretion No requirement for drugs affecting bone marrow function (e.g., lithium, corticosteroids) No medical condition precluding postoperative chemotherapy No prior or concurrent malignancy other than nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior locoregional radiotherapy to the head and neck Surgery: Excision with curative intent required

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 1994-02; Primary Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bernier, MD, PhD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (19):
- Institut Jules Bordet, Brussels, Belgium
- France (6):
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Oscar Lambret, Lille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Hopital Jean Bernard, Poitiers
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- University Medical Center Nijmegen, Nijmegen, Netherlands
- Medical University of Gdansk, Gdansk, Poland
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Ciudad Sanitaria Vall D'Hebron, Barcelona, Spain
- Switzerland (4):
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitaetsspital, Zurich
- Dokuz Eylul University School of Medicine, Izmir, Turkey (Türkiye)
- Nottingham City Hospital NHS Trust, Nottingham, England, United Kingdom

REFERENCES:
- [Result] Bernier J, Cooper JS, Pajak TF, van Glabbeke M, Bourhis J, Forastiere A, Ozsahin EM, Jacobs JR, Jassem J, Ang KK, Lefebvre JL. Defining risk levels in locally advanced head and neck cancers: a comparative analysis of concurrent postoperative radiation plus chemotherapy trials of the EORTC (#22931) and RTOG (# 9501). Head Neck. 2005 Oct;27(10):843-50. doi: 10.1002/hed.20279. PMID 16161069
- [Result] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Result] Bernier J, Domenge C, Eschwege F, et al.: Chemo-radiotherapy, as compared to radiotherapy alone, significantly increases disease-free and overall survival in head and neck cancer patients after surgery: results of EORTC phase III trial 22931. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-1, 1, 2001.
- [Result] Valley JF, Bernier J, Tercier PA, Fogliata-Cozzi A, Rosset A, Garavaglia G, Mirimanoff RO. Quality assurance of the EORTC radiotherapy trial 22931 for head and neck carcinomas: the dummy run. Radiother Oncol. 1998 Apr;47(1):37-44. doi: 10.1016/s0167-8140(97)00218-1. PMID 9632290